CLINICAL TRIAL: NCT05125250
Title: Effects of Vestibular Exercises and Motor Control on Cervical Spine Range of Motion and Balance in Cervicogenic Dizziness
Brief Title: Effects of Vestibular Exercises and Motor Control in Cervicogenic Dizziness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/00963 Amber
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Control Group (Experimental): This group will receive treatment which comprises of therapeutic exercises, During the first 4 weeks, motor control and ROM exercises will be prescribed in order to improve muscular endurance of deep flexors muscles and to improve the ROM of cervical spine in flexion, extension, rotation and side bending and lateral rotation in. These exercises will be performed at a rate of 3 sets and an intensity of 15 repetitions per day
  Interventions: Other: Motor Control Group
- Vestibular Group (Active Comparator): This Group will receive vestibular exercises which comprises of postural awareness training; Standing on a balance board, Foveal vision exercises.
  Interventions: Other: Vestibular Group

INTERVENTIONS:
Other: Motor Control Group — will received treatment which comprises of therapeutic exercises, During the first 4 weeks, motor control and ROM exercises will be prescribed in order to improve muscular endurance of deep flexors muscles and to improve the ROM of cervical spine in flexion, extension, rotation and side bending and lateral rotation in. These exercises will be performed at a rate of 3 sets and an intensity of 15 repetitions per day .
  Arms: Motor Control Group
Other: Vestibular Group — will receive vestibular exercises which comprises of postural awareness training, balance board exercises, Foveal vision exercises .
  Arms: Vestibular Group

SUMMARY:
The feelings of imbalance, unsteadiness, and disorientation with cervicogenic dizziness is not clear. It has been suggested that a disruption of the normal afferent signals from the upper cervical proprioceptors to the vestibular nucleus results in an inaccurate depiction of head and neck orientation in space due to highly developed proprioceptive system that allows the neuromuscular control of cervical spine and effective use of vital organs in the head through unique connections to the vestibular and visual systems. Motor Control Therapeutic Exercises and vestibular exercises have been used to increase motor control and reduce pain and disability in patients with neck pain.

DETAILED DESCRIPTION:
Cervicogenic dizziness is defined as a sensation of instability or disequilibrium that occurs with the pain and stiffness in cervical spine and is aggravated by neck movements or positions. Dizziness is a common indication in people with cervical spine dysfunction. cervicogenic dizziness as "a nonspecific sensation of altered orientation in space and disequilibrium originating from abnormal afferent activity from the neck" which is thought to be caused by disorders in the upper cervical spine and commonly it is associated with cervical stiffness neck pain or headache.

Motor control can also be defined as the capacity of how the central nervous system produces of useful movements that are coordinated and integrated with the rest of the body and the environment. Thus, motor control therapeutic exercises (MCTE) are used to improve the conditions of patients. Motor Control Therapeutic Exercises have been used to increase motor control and reduce pain and disability in patients with neck pain. MCTE comprised of cranio-cervical flexor exercise, cranio-cervical extensor exercise, co-contraction of flexors and extensors, a synergy exercise for retraining the strength of the deep neck flexors.

Schenk et al. have published case studies in which they describe the diagnosis, treatment, and outcomes of a patient with cervicogenic dizziness co-managed by a vestibular and an orthopedic manual physical therapist. They argue that manual therapy combined with vestibular rehabilitation may be superior in the treatment of cervicogenic dizziness. Literature states that vestibular exercises have been used to increase motor control and reduce pain and disability in patients with neck pain.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 30-65 years

  * Gender both
  * Pain and dizziness lasting for at least 3 months;
  * Pain intensity corresponding to at least 3 points on a 10-point numeric pain rating scale;
  * Restricted cervical range of movement (flexion, extension, rotation and side-bending);
  * Presence of neck pain associated with disability according to the NDI greater than or equal to 5 points;
  * Presence of subjective dizziness associated with pain, movement, stiffness or specific postures of the cervical region

Exclusion Criteria:

* • Any other systemic or neurodegenerative pathology, presence of trauma or recent surgery to the head, face, neck or chest;

  * specific diagnosis of central or peripheral dizziness;
  * History of previous physical-therapy intervention for the cervical region;
  * Any cognitive impairment that hindered viewing of audiovisual material;
  * Difficulty understanding or communicating

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory Scale | Change from Baseline ,dizziness to 4Weeks, 8 weeks
  The purpose of this scale is to identify difficulties that you may be experiencing because of your dizziness. It has three subscales namely physical, emotional and functional. The total maximum score is 100 and minimum is 0.
Neck Disability Index (NDI) | Change from Baseline , to 4Weeks, 8 weeks
  This questionnaire has been designed to give us information as to how your neck pain has affected your ability to manage in everyday life. Is 10 item scale each item assesses different neck pain complaints. The total maximum score is 50 and minimum is 0
Berg Balance Scale | Change from Baseline , balance and fall prevention to 4Weeks, 8 weeks
  Berg Balance Scale is a 14 items scale, to assess static and dynamic balance. Scoring of this scale is done on a 5 point scale where 0 is inability to perform a task and 4 shows the independent task performance. The maximum score of this scale is 56 showing excellent performance

CONTACTS AND LOCATIONS:
Overall Officials: Misbah Ghous, Principal Investigator — Riphah college of Rehabilitation and Allied Health sciences Islamabad
Locations (1):
- Pakistan General Railway Hospital, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lystad RP, Bell G, Bonnevie-Svendsen M, Carter CV. Manual therapy with and without vestibular rehabilitation for cervicogenic dizziness: a systematic review. Chiropr Man Therap. 2011 Sep 18;19(1):21. doi: 10.1186/2045-709X-19-21. PMID 21923933
- [Background] 4. Schenk RP, Coons LB, Bennett SE, Huijbregts PA. Cervicogenic dizziness: a case report illustrating orthopaedic manual and vestibular physical therapy comanagement. Journal of Manual & Manipulative Therapy. 2006 Jul 1;14(3):56E-68E.
- [Background] Schenk R, Coons LB, Bennett SE, Huijbregts PA: Cervicogenic dizziness: A case report illustrating manual and vestibular physical therapy comanagement. The Journal of Manual & Manipulative Therapy. 2006, 14 (3): E56-E68.